CLINICAL TRIAL: NCT00311662
Title: Multi-centre, Parallel Group, Double-blind, Placebo Controlled Study of the Efficacy and Tolerability of Tonabersat in the Prophylaxis of Migraine Headache
Brief Title: Efficacy and Tolerability of Tonabersat in the Prophylaxis of Migraine Headache
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Minster Research Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TON/01/05-CLIN
Record Dates: First submitted 2006-04-04; First posted 2006-04-06 (Estimated); Last update posted 2009-08-31 (Estimated); Status verified 2009-08

CONDITIONS: Migraine Without Aura; Migraine With Aura
MeSH Terms: conditions — Migraine without Aura; Migraine with Aura | interventions — tonabersat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Tonabersat 40mg
  Interventions: Drug: Tonabersat
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tonabersat — Tablet 40mg daily for 12 weeks
  Other Names: SB220453
  Arms: 1
Drug: Placebo — Tablet once daily for 12 weeks
  Arms: 2

SUMMARY:
Overall trial objectives:

* Can treatment with tonabersat reduce the number of days with a migraine headache in patients who suffer from frequent migraine attacks
* How well tolerated is treatment with tonabersat

The study is based on the hypothesis that the unique mechanism of action of tonabersat will inhibit some of the early events in the generation of migraine and so be effective as prophylactic treatment

ELIGIBILITY:
Inclusion Criteria:

* An established history of migraine of at least one year, with or without aura, meeting the diagnostic criteria of the International Classification of Headache Disorders, and experience between four and 14 migraine headache days per month; headache days should be experienced within at least two and no more than six migraine attacks per month.
* Women of child bearing potential must be using a reliable form of contraception (defined in the protocol) for at least three months prior to enrolment with contraception maintained for at least 7 days after the last dose of study medication and they must have a negative pregnancy test at screening with no intention of becoming pregnant during the study period.

Exclusion Criteria:

* Patients with a diagnosis of migraine according to the diagnostic criteria of the International Classification of Headache Disorders at age 50 years or more.
* Experience frequent non-migraine headache
* Patients with pure menstrual migraine defined as patients in whom migraine attacks occur exclusively on Day 1 +/- 2 (i.e. Days -2 to +3) of menstruation in at least two out of three menstrual cycles and at no other times of the cycle.
* Patients with other significant central nervous system disorders in the opinion of the investigator.
* Failure to respond to more than two adequately dosed (i.e. recommended total daily dose and of sufficient duration) migraine prophylactic medications.
* Overuse of acute migraine treatments defined as more than 14 medication days per month with analgesics and opioids and nine medication days per month of ergots or triptans.
* Prophylactic treatment within two months prior to entry to the trial.
* Patients taking any of the following medications: beta-blockers (during the last two months), tricyclic antidepressants (during the last two months), antiepileptic drugs (during the last two months), calcium channel blockers (during the last two months), monoamine oxidase inhibitors (during the last two months), daily oral NSAIDs, daily paracetamol, high dose magnesium supplements (600 mg/day), daily multivitamin preparations containing more than 10 mg riboflavin, daily use of oral corticosteroids and daily herbal preparations (e.g. feverfew, butterwort and St John's Wort). Parenteral administration of Botulinum toxin is also excluded. Patients taking other medications used as prophylaxis for migraine including methysergide, anti spasticity agents (e.g. tizanidine) and the new generation antipsychotics (e.g. olanzapine) currently or within the previous two months should also be excluded.
* Patients who, in the opinion of the investigator, have significant cerebrovascular disease, e.g. transient ischaemic attacks, stroke.
* Patients who, in the opinion of the investigator, have clinically significant cardiovascular disease.
* Patients suffering from a current clinical diagnosis of major depressive disorder or schizophrenia.
* Patients with renal dysfunction, defined as a serum creatinine of greater than 125% of the upper limit of normal for their age group.
* Patients with hepatic dysfunction defined as a liver function test (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase, bilirubin) of greater than twice the upper limit of normal for their age group.
* Patients with known alcohol or other substance abuse.
* Failure to complete the diary card during the baseline period.
* Participation in another clinical trial in the previous four weeks.
* Any women who is pregnant, lactating or not using medically acceptable contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2006-04; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Change in the mean monthly number of migraine headache days from the baseline period to Month 3. | weeks 8 to 12 compared to weeks -4 to 0
Incidence of all adverse events (AEs), serious AEs and AEs leading to withdrawal of trial medication, clinical laboratory tests, vital signs and physical examination | 12 weeks

SECONDARY OUTCOMES:
Change in the mean monthly number of migraine headache days from the baseline period to across the whole treatment period. | weeks 0-12 compared to weeks -4 to 0
Proportion of patients defined as a responder, i.e. those with a reduction of at least 50% in the mean monthly number of migraine headache days in the third month of treatment and over the whole treatment period. | weeks 8-12 compared to weeks -4 to 0
Change in mean monthly number of migraine attacks from the baseline period to Month 3. | weeks 8-12 compared to weeks -4 to 0
Change in mean monthly number of migraine attacks from the baseline period to across the whole treatment period. | weeks 0 to 12 compared to weeks -4 to 0
Proportion of patients defined as a responder, i.e. those with a reduction of at least 50% in the mean monthly frequency of migraine attacks in the third month of treatment and over the whole treatment period. | weeks 8-12 compared to weeks -4 to 0
Speed of effect of treatment. | 12 weeks
Change in the mean monthly consumption of rescue medication from the baseline period to Month 3. | weeks 8 to 12 compared to weeks -4 to 0
Change in the mean monthly consumption of rescue medication from the baseline period to across the whole treatment period. | weeks 0 to 12 comoared to weeks -4 to 0
Overall severity of migraine attacks occurring during the treatment period. | 12 weeks
Overall response to the question "How satisfied are you with the trial medication?" | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Goadsby, MD, Principal Investigator — The National Hospital for Neurology and Neurosurgery, London
Locations (17):
- Denmark (2):
  - Glostrup Amtssygehus, Neurologisk Ambulatorium N01, Copenhagen
  - Bispebjerg Hospital, Neurolgisk Afdeling N, Copenhagen
- Hungary (4):
  - Kenézy Gyula County Hospital, Dept of Neurology, Debrecen
  - Petz Aladár Megyei Oktató Kórház, Győr
  - Borsod Abauj Zemplén Megyei Kórház, Neurologiai Osztaly, Miskolc
  - Zala County Hospital, Department of Cardiology, Zalaegerszeg
- South Africa (10):
  - Quinta-Med, Bloemfontein
  - Chris Barnard Memorial Hospital, Cape Town
  - St. Augustine's Medical Mews, Durban
  - Francois Le Clus, Johannesburg
  - Dr I Engelbrecht, Lyttleton
  - Pretoria East Hospital, Neuro-Orthopaedic Unit, Pretoria
  - Intercare Corporate Office, Pretoria
  - Dr J Bouwer, Pretoria
  - Little Company of Mary, Neurospinal Building, Pretoria
  - SCION Clinical Research, 316 Medi-Clinic Heart Hospital, Pretoria
- The National Hospital for Neurology & Neurosurgery, London, United Kingdom

REFERENCES:
- [Background] Tfelt-Hansen P, Block G, Dahlof C, Diener HC, Ferrari MD, Goadsby PJ, Guidetti V, Jones B, Lipton RB, Massiou H, Meinert C, Sandrini G, Steiner T, Winter PB; International Headache Society Clinical Trials Subcommittee. Guidelines for controlled trials of drugs in migraine: second edition. Cephalalgia. 2000 Nov;20(9):765-86. doi: 10.1046/j.1468-2982.2000.00117.x. No abstract available. PMID 11167908
- [Background] Lauritzen M. Pathophysiology of the migraine aura. The spreading depression theory. Brain. 1994 Feb;117 ( Pt 1):199-210. doi: 10.1093/brain/117.1.199. PMID 7908596
- [Background] Committee for Proprietary Medicinal Products. Note for guidance on clinical investigation of medicinal products for the treatment of migraine, CPMP/EWP/788/01/Final. London, 17 December 2003.
- [Result] Goadsby PJ, Ferrari MD, Csanyi A, Olesen J, Mills JG; Tonabersat TON-01-05 Study Group. Randomized, double-blind, placebo-controlled, proof-of-concept study of the cortical spreading depression inhibiting agent tonabersat in migraine prophylaxis. Cephalalgia. 2009 Jul;29(7):742-50. doi: 10.1111/j.1468-2982.2008.01804.x. Epub 2009 Feb 13. PMID 19222510